CLINICAL TRIAL: NCT06389188
Title: Effectiveness of Cervical Osteopathic Manipulation Techniques of High Velocity and Low Amplitude in Patients with Whiplash- Associated Disorders
Brief Title: Effectiveness of Cervical Osteopathic Manipulation in Patients with Whiplash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, JOSE VICENTE TOLEDO MARHUENDA, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JVT003
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-05

CONDITIONS: Whiplash
Keywords: manual therapy; manipulation; physical therapy; exercises
MeSH Terms: conditions — Whiplash Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: MAN Group (Experimental): MAN-Group were treated with cervical spine manipulation with SAT. Patients received a total of 3 sessions of treatment over a month (days 1, 15 and 30 after the beginning of the study).
  Interventions: Procedure: RHB Group
- MAN Group (Active Comparator): MAN-Group were treated with cervical spine manipulation with SAT. Patients received a total of 3 sessions of treatment over a month (days 1, 15 and 30 after the beginning of the study).
  Interventions: Procedure: RHB Group

INTERVENTIONS:
Procedure: RHB Group — The RHB-group were treated with passive manual therapy (P-MT) by soft tissue mobilization, massage and muscular stretching of the anterior and posterior cervical muscles; active therapeutic exercises (A-TE); and oculo-cervical exercises (OC-E). Patients received a total of 20 sessions of 30 minutes each during 4 weeks

SUMMARY:
To determine the mid- and long-term efficiency (15, 30 and 120 days after starting sessions) of the SAT technique in patients with grade II acute WL, comparing it with a conventional rehabilitation program.

DETAILED DESCRIPTION:
A prospective, single-blind, parallel group, randomized, will be carried out in the physiotherapy service of the Clinic Hospital of Terrassa with the participation of the rehabilitation, radiology, traumatology and surgery services.

Patients will be recruited from emergency services of the Clinic Hospital of Terrassa and randomly divided into two groups MAN-Group and RHB-Group, using the random number generator of a statistical program (SPSS), to receive 3 and 20 treatment sessions, respectively.

The treatment protocol was carried out during four weeks, and both interventions occurred over the same time period. In both treatment groups, patients started sessions during the first two week after the traffic car collision.

MAN-Group were treated with cervical spine manipulation with SAT, after specialized physical therapists assessed there was no risk of vertebro-basilar injuries following the International Framework. Patients received a total of 3 sessions of treatment over a month (days 1, 15 and 30 after the beginning of the study).

The RHB-group were treated with passive manual therapy (P-MT) by soft tissue mobilization, massage and muscular stretching of the anterior and posterior cervical muscles; active therapeutic exercises (A-TE); and oculo-cervical exercises (OC-E). Patients received a total of 20 sessions of 30 minutes each during 4 weeks. The exercises were performed five times (30 seconds interval each time) in a sitting position.

ELIGIBILITY:
Inclusion Criteria:

Patients between 18-60 years of age Who went to the emergency service after suffering a traffic car collision being the driver of the car.

With acute WL grade II WAD diagnosis, made by physicians from the traumatology service (with neck pain by whiplash trauma with objective findings but no radiculopathy).

Referred to the hospital rehabilitation service

Exclusion Criteria:

Any other symptomatology different to neck pain and other coexisting medical conditions which could severely restrict participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Subjective pain intensity | At baseline and at week 2, 4 and follow-up.
  Neck pain intensity was assessed with a Visual Analogue Scale (VAS) to measure the amount of pain experienced by a subject from both groups on a continuum from 0 to 100 mm. Scores can range from 0 (no pain) to 100 (worst imaginable pain)19,20. This method has been proven to be a reliable, generalizable and internally consistent measure of clinical and experimental neck pain
Neck specific disability | At baseline and at week 2, 4 and follow-up.
  Neck-specific disability was measured with Neck Disability Index (NDI). The NDI is a valid measurement of disability in neck pain disorders. It is widely used and it has shown good reliability and validity in WAD studies. NDI scores can range from 0% (no limitation on activity) to 100% (worst possible disability).

SECONDARY OUTCOMES:
Cervical range of motion (CROM) | At baseline and at week 2 and week 4.
  Neck range of motion was tested with the CROM Instrument. All cervical motions and subsequent measurements were performed according to the manufacturer's specifications and were reproduced exactly for each trial with a single examiner performing all measurements. CROM were assessed in a relaxed sitting position, hips and knees positioned at 90º angles and buttocks positioned against the back of the chair. The goniometer was placed on the top of the head and was set in the neutral position.
Cervical lordosis Cobb angle | At baseline and at week 4.
  Cobb angle (COBB) method was measured to assess cervical lordosis (Cobb C2-C7) as the angle between the horizontal line on the lower endplate of C2 and a horizontal line on the lower endplate of C7. A clinically normal cervical lordosis has been described as a Cobb angle of 31-40 degrees, with subjects in standing and eyes focused straight ahead. A cervical lordosis of less than 20◦ from C2 to C7 has been shown to be related to cervical dysfunction and pain.
Hospital anxiety and depression scale | At baseline and at week 4 and follow-up.
  HADS was used to determine the levels of anxiety and depression experienced by participants. HADS has 14 items and it was designed for the evaluation of anxiety and depression in non-psychiatric outpatient hospital services. The entire sum for both HADS anxiety and HADS depression levels ranges from 0 to 21. A score equal to or more than 10 indicates clinically significant symptoms of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Parera-Turull, PhD., Principal Investigator — Clinical Research Centre d'Osteopatia Terrassa. Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa., Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peolsson A, Landen Ludvigsson M, Tigerfors AM, Peterson G. Effects of Neck-Specific Exercises Compared to Waiting List for Individuals With Chronic Whiplash-Associated Disorders: A Prospective, Randomized Controlled Study. Arch Phys Med Rehabil. 2016 Feb;97(2):189-95. doi: 10.1016/j.apmr.2015.10.087. Epub 2015 Oct 26. PMID 26514296
- [Background] De Rosario H, Vivas MJ, Sinovas MI, Page A. Relationship between neck motion and self-reported pain in patients with whiplash associated disorders during the acute phase. Musculoskelet Sci Pract. 2018 Dec;38:23-29. doi: 10.1016/j.msksp.2018.09.004. Epub 2018 Sep 6. PMID 30218881
- [Background] Rasmussen C, Stenager E, Nielsen CV. [Social, economic and cultural aspects of whiplash syndrome]. Ugeskr Laeger. 2010 Jun 14;172(24):1815-7. Danish. PMID 20566153
- [Background] Walton DM, Elliott JM. An Integrated Model of Chronic Whiplash-Associated Disorder. J Orthop Sports Phys Ther. 2017 Jul;47(7):462-471. doi: 10.2519/jospt.2017.7455. Epub 2017 Jun 16. PMID 28622487
- [Background] Spitzer WO, Skovron ML, Salmi LR, Cassidy JD, Duranceau J, Suissa S, Zeiss E. Scientific monograph of the Quebec Task Force on Whiplash-Associated Disorders: redefining "whiplash" and its management. Spine (Phila Pa 1976). 1995 Apr 15;20(8 Suppl):1S-73S. No abstract available. PMID 7604354
- [Background] Wiangkham T, Duda J, Haque S, Madi M, Rushton A. The Effectiveness of Conservative Management for Acute Whiplash Associated Disorder (WAD) II: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. PLoS One. 2015 Jul 21;10(7):e0133415. doi: 10.1371/journal.pone.0133415. eCollection 2015. PMID 26196127
- [Background] 7. Regal Ramos, R.J. Síndrome de latigazo cervical: Características epidemiológicas de los pacientes evaluados en la unidad médica de valoración de incapacidades de Madrid. Medicina y Seguridad del Trabajo 225:348-360 (2011).
- [Background] Pajediene E, Janusauskaite J, Samusyte G, Stasaitis K, Petrikonis K, Bileviciute-Ljungar I. Patterns of acute whiplash-associated disorder in the Lithuanian population after road traffic accidents. J Rehabil Med. 2015 Jan;47(1):52-7. doi: 10.2340/16501977-1892. PMID 25315016
- [Background] Peolsson A, Landen Ludvigsson M, Peterson G. Neck-specific exercises with internet-based support compared to neck-specific exercises at a physiotherapy clinic for chronic whiplash-associated disorders: study protocol of a randomized controlled multicentre trial. BMC Musculoskelet Disord. 2017 Dec 12;18(1):524. doi: 10.1186/s12891-017-1853-1. PMID 29233141
- [Background] Peterson G, Dedering A, Andersson E, Nilsson D, Trygg J, Peolsson M, Wallman T, Peolsson A. Altered ventral neck muscle deformation for individuals with whiplash associated disorder compared to healthy controls - a case-control ultrasound study. Man Ther. 2015 Apr;20(2):319-27. doi: 10.1016/j.math.2014.10.006. Epub 2014 Oct 15. PMID 25454684
- [Background] Peolsson A, Karlsson A, Ghafouri B, Ebbers T, Engstrom M, Jonsson M, Wahlen K, Romu T, Borga M, Kristjansson E, Bahat HS, German D, Zsigmond P, Peterson G. Pathophysiology behind prolonged whiplash associated disorders: study protocol for an experimental study. BMC Musculoskelet Disord. 2019 Feb 2;20(1):51. doi: 10.1186/s12891-019-2433-3. PMID 30711003
- [Background] Elkin BS, Elliott JM, Siegmund GP. Whiplash Injury or Concussion? A Possible Biomechanical Explanation for Concussion Symptoms in Some Individuals Following a Rear-End Collision. J Orthop Sports Phys Ther. 2016 Oct;46(10):874-885. doi: 10.2519/jospt.2016.7049. PMID 27690834
- [Background] Church EW, Sieg EP, Zalatimo O, Hussain NS, Glantz M, Harbaugh RE. Systematic Review and Meta-analysis of Chiropractic Care and Cervical Artery Dissection: No Evidence for Causation. Cureus. 2016 Feb 16;8(2):e498. doi: 10.7759/cureus.498. PMID 27014532
- [Background] Haldeman S, Carroll L, Cassidy JD, Schubert J, Nygren A. The Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders: executive summary. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S7-9. doi: 10.1016/j.jmpt.2008.11.005. No abstract available. PMID 19251077
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL; COG. Manipulation or mobilisation for neck pain: a Cochrane Review. Man Ther. 2010 Aug;15(4):315-33. doi: 10.1016/j.math.2010.04.002. Epub 2010 May 26. PMID 20510644